CLINICAL TRIAL: NCT01004237
Title: Additive Effects of Pravastatin and Valsartan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Dr. Koh, Gachon University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GMC-200912
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2010-10

CONDITIONS: Hypertension; High Cholesterol
Keywords: insulin resistance; hypertensive; hypercholesterolemic patients
MeSH Terms: conditions — Hypertension; Hypercholesterolemia; Insulin Resistance | interventions — Pravastatin; Valsartan

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- pravastatin (Active Comparator)
  Interventions: Drug: pravastatin, valsartan, pravastatin+valsartan
- valsartan (Active Comparator)
  Interventions: Drug: pravastatin, valsartan, pravastatin+valsartan
- pravastatin combined with valsartan (Active Comparator)
  Interventions: Drug: pravastatin, valsartan, pravastatin+valsartan

INTERVENTIONS:
Drug: pravastatin, valsartan, pravastatin+valsartan — pravastatin 40 mg, valsartan 160 mg 8 weeks of treatment

SUMMARY:
The investigators hypothesize that pravastatin combined with valsartan may have additive effects in hypertensive, hypercholesterolemic patients.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension and low-density lipoprotein cholesterol levels >100

Exclusion Criteria:

* Overt liver disease Chronic renal failure Hypothyroidism Myopathy Uncontrolled diabetes Severe hypertension

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
flow-mediated dilation | 8 weeks of treatment

SECONDARY OUTCOMES:
insulin resistance | 8 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Gil Medical Center, Incheon, South Korea

REFERENCES:
- [Derived] Koh KK, Lim S, Choi H, Lee Y, Han SH, Lee K, Oh PC, Sakuma I, Shin EK, Quon MJ. Combination pravastatin and valsartan treatment has additive beneficial effects to simultaneously improve both metabolic and cardiovascular phenotypes beyond that of monotherapy with either drug in patients with primary hypercholesterolemia. Diabetes. 2013 Oct;62(10):3547-52. doi: 10.2337/db13-0566. Epub 2013 Jul 17. PMID 23863812